CLINICAL TRIAL: NCT02538588
Title: Comparison of Amikacin Lung Delivery With Two Nebulizers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Akeflow
Record Dates: First submitted 2015-08-24; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Healthy; Cystic Fibrosis
Keywords: Healthy Volunteers
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebulizer 1 (Experimental): Nebulization with akita nebulizer
  Interventions: Device: Nebulizer 1
- Nebulizer 2 (Active Comparator): Nebulization with eFlow nebulizer
  Interventions: Device: Nebulizer 2

INTERVENTIONS:
Device: Nebulizer 1
  Other Names: Akita
  Arms: Nebulizer 1
Device: Nebulizer 2
  Other Names: eFlow
  Arms: Nebulizer 2

SUMMARY:
Comparison between two modalities of nebulization.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy subjects
* Cystic fibrosis

Exclusion Criteria:

* Kidney failure
* No pregnancy

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Total urinary concentration of amikacin | 24 hours after the nebulization
  Pharmacokinetic study of the urinary excretion of amikacin after nebulization

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium